CLINICAL TRIAL: NCT06807424
Title: A Phase 3, Multicenter, Randomized, Double-blind, Placebo-controlled Study Evaluating the Efficacy and Safety of JNJ-77242113 for the Treatment of Biologic-experienced Participants With Active Psoriatic Arthritis
Brief Title: A Study to Evaluate the Efficacy and Safety of Icotrokinra (JNJ-77242113) in Biologic-experienced Participants With Active Psoriatic Arthritis
Acronym: ICONIC-PsA 2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77242113PSA3002; 77242113PSA3002 (Other: Janssen Research & Development, LLC); 2024-517284-23-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Psoriatic
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I: Icotrokinra Dose 1 (Experimental): Participants will receive icotrokinra Dose 1. Participants who have not discontinued will be eligible to enter a long term extension (LTE) and will continue to receive icotrokinra Dose 1.
  Interventions: Drug: Icotrokinra
- Group II: Icotrokinra Dose 2 (Experimental): Participants will receive icotrokinra Dose 2. Participants who have not discontinued will be eligible to enter a LTE and will continue to receive icotrokinra Dose 2.
  Interventions: Drug: Icotrokinra
- Group III: Placebo (Placebo Comparator): Participants will receive placebo matched to icotrokinra and will cross over to receive icotrokinra Dose 1 or Dose 2 at Week 16. Participants who have not discontinued will be eligible to enter a LTE and will continue to receive icotrokinra Dose 1 or Dose 2.
  Interventions: Drug: Icotrokinra; Drug: Placebo

INTERVENTIONS:
Drug: Icotrokinra — Icotrokinra will be administered.
  Other Names: JNJ-77242113
Drug: Placebo — Placebo will be administered.
  Arms: Group III: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of icotrokinra compared to placebo in biologic-experienced participants with active psoriatic arthritis (PsA) by assessing the reduction in signs and symptoms of PsA.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have been previously treated with 1 biologic agent for psoriatic arthritis (PsA) or psoriasis and have discontinued treatment for any reason. The reason for discontinuation must be documented
* Have a diagnosis of psoriatic arthritis (PsA) for at least 3 months before the first administration of study intervention and meet classification criteria for Psoriatic Arthritis (CASPAR) at screening
* Have active PsA as defined by: (a) At least 3 swollen joints and at least 3 tender joints at screening and at baseline (b) C-reactive protein (CRP) greater than or equal to (>=) 0.1 milligrams per deciliter (mg/dL) at screening from the central laboratory
* Have at least 1 of the PsA subsets: distal interphalangeal joint involvement, polyarticular arthritis with absence of rheumatoid nodules, arthritis mutilans, asymmetric peripheral arthritis, or spondylitis with peripheral arthritis
* Have active plaque psoriasis with at least one psoriatic plaque of >= 2 cm diameter or nail changes consistent with psoriasis
* A female participant of childbearing potential must have a negative highly sensitive serum pregnancy test (Beta-hCG) at screening and a negative urine pregnancy test at Week 0 prior to administration of study intervention

Exclusion Criteria:

* Has a history or current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic (with the exception of PsA), psychiatric, genitourinary, or metabolic disturbances
* Currently has a malignancy or has a history of malignancy within 5 years prior to screening
* Has known allergies, hypersensitivity, or intolerance to icotrokinra or its excipients
* Has other inflammatory diseases that might confound the evaluations of benefit of icotrokinra therapy, including but not limited to rheumatoid arthritis (RA), systemic lupus erythematosus, or Lyme disease
* Participants with fibromyalgia or osteoarthritis symptoms that, in the investigator's opinion, would have potential to interfere with efficacy assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2025-01-09 (Actual); Primary Completion 2027-02-10 (Estimated); Study Completion 2028-10-18 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants who Achieved an American College of Rheumatology (ACR) 20 Response at Week 16 | Week 16
  The ACR 20 responders are participants with an improvement of greater than or equal to (>=) 20 percent (%) from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain visual analog scale (VAS), patient's global assessment of disease activity [arthritis, VAS] scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein).

SECONDARY OUTCOMES:
Proportion of Participants Who Achieved Psoriatic Area and Severity Index (PASI) 75 Response at Week 16 Among Participants with Baseline Body Surface Area (BSA) Greater Than Equal to (>=) 3 Percent (%) and With Baseline IGA Score of >=2 | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 75 response represents participants who achieved at least a 75 percent improvement from baseline in the PASI score.
Proportion of Participants Who Achieved PASI 90 Response at Week 16 Among Participants with Baseline BSA >=3% and With Baseline IGA Score of >=2 | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 90 response represents participants who achieved at least a 90 percent improvement from baseline in the PASI score.
Proportion of Participants Who Achieved PASI 100 Response at Week 16 Among Participants with Baseline BSA >=3% and With Baseline IGA Score of >=2 | Week 16
  The PASI is a system used for assessing and grading the severity of psoriatic lesions. In the PASI system, the body is divided into 4 regions: the head, trunk, upper extremities, and lower extremities. Each of these areas were assessed separately for the percentage of the area involved, which translates to a numeric score that ranges from 0 to 6, and for erythema, induration, and scaling, which are each rated on a scale of 0 to 4. The PASI produces a numeric score that can range from 0 to 72. A higher score indicates more severe disease. A PASI 100 response represents participants who achieved at least a 100 percent improvement from baseline in the PASI score.
Proportion of Participants with an Investigator Global Assessment (IGA) Psoriasis Score of 0 or 1 And >=2 Grade Improvement From Baseline at Week 16 Among Participants with Baseline BSA >=3% and With Baseline IGA Score of >=2 | Week 16
  Proportion of participants with an IGA psoriasis score of 0 or 1 And >=2 grade improvement from baseline at Week 16 among participants with >=3% BSA and an IGA Score of >=2 at Baseline will be reported. The IGA documents the investigator's assessment of the participant's psoriasis at a given time point. Overall lesions are graded for induration, erythema, and scaling, each using a 5-point scale: using 0 (no evidence), 1 (minimal), 2 (mild), 3 (moderate), and 4 (severe) scale. The IGA score of psoriasis is based upon the average of induration, erythema, and scaling scores. The participant's psoriasis is assessed as cleared (0), minimal (1), mild (2), moderate (3), or severe (4).
Proportion of Participants who Achieved an ACR 50 Response at Week 16 | Week 16
  The ACR 50 responders are participants with an improvement of >= 50% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity (arthritis, VAS) scale, Physician's global assessment of disease activity VAS scale, Health Assessment Questionnaire and C-reactive protein).
Proportion of Participants who Achieved an ACR 70 Response at Week 16 | Week 16
  The ACR 70 responders are participants with an improvement of >= 70% from baseline in both the tender and swollen joint count and in at least 3 of the 5 assessments (patient's assessment of pain VAS, patient's global assessment of disease activity (arthritis, VAS) scale, Physician's global assessment of disease activity VAS scale, health assessment questionnaire and C-reactive protein).
Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score At Week 16 | From baseline up to Week 16
  The HAQ-DI score consists of questions referring to 8 categories: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and common daily activities. Responses in each functional area are scored from 0 to 3 (0=no difficulty and 3=inability to perform a task in that area). Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Changes From Baseline in 36 Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 16 | From baseline up to Week 16
  SF-36 is a standardized survey evaluating 8 aspects of functional health and wellbeing: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a domain was an average of the individual question scores, which were scaled 0 to 100 (100=highest level of functioning). Score from physical function, role physical, bodily pain, and general health domains were averaged to calculate PCS. Total score range for PCS was 0-100 (100=highest level of physical functioning).
Proportion of Participants With Resolution of Enthesitis at Week 16 Among Those With Enthesitis at Baseline | Week 16
  Enthesitis will be assessed using the Leeds Enthesitis Index (LEI). The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Change From Baseline in Enthesitis Score at Week 16 in Participants With Enthesitis at Baseline | Baseline and Week 16
  Enthesitis will be assessed using the LEI. The LEI was developed to assess enthesitis in participants with PsA, and evaluates the presence (score of 1) or absence of pain (score of 0) by applying local pressure to Lateral elbow epicondyle, left and right, Medial femoral condyle, left and right, and Achilles tendon insertion, left and right. LEI scores ranging from 0 (0 sites with tenderness) to 6 (worst possible score; 6 sites with tenderness).
Proportion of Participants With Resolution of Dactylitis at Week 16 Among Those With Dactylitis at Baseline | Week 16
  Dactylitis is characterized by swelling of the entire finger or toe. Presence and severity of dactylitis will be assessed in both hand and feet using a scoring system from 0 to 3 (0: no dactylitis, 1: mild dactylitis, 2: moderate dactylitis, 3: severe dactylitis). The result for each digit are summed to produce a final dactylitis score with a range from 0 to 60. Higher score indicates greater severity.
Change From Baseline in Dactylitis Score at Week 16 in Participants With Dactylitis at Baseline | From baseline up to Week 16
  Dactylitis is characterized by swelling of the entire finger or toe. Presence and severity of dactylitis will be assessed in both hand and feet using a scoring system from 0 to 3 (0: no dactylitis, 1: mild dactylitis, 2: moderate dactylitis, 3: severe dactylitis). The result for each digit are summed to produce a final dactylitis score with a range from 0 to 60. Change from baseline in dactylitis score measure the change in dactylitis, where a negative change indicates an improvement and a positive change indicates a worsening.
Proportion of Participants who Achieved Minimal Disease Activity (MDA) at Week 16 | Week 16
  MDA criteria are a composite of 7 outcome measures used in PsA. Participants are classified as achieving MDA if they fulfill at least 5 out of the 7 outcome measures: tender joint count less than or equal to (<=) 1; swollen joint count <= 1; psoriasis activity and severity index <= 1 or body surface area <= 3 percent (%); patient pain VAS score of <= 15; patient global disease activity VAS (arthritis and psoriasis) score of <= 20; health assessment questionnaire (HAQ) score <= 0.5; and tender entheseal points <= 1.
Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 16 | From baseline up to Week 16
  The FACIT-fatigue is a self-administered, 13 item questionnaire measuring items on tiredness, weakness, and difficulty conducting usual activities due to fatigue. Responses to all items are rated on a 5-point Likert response scale ranging from 0 "not at all" to 4 "very much." The total score ranges from 0 to 52, with higher values indicating less fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (214):
- United States (23):
  - AARA Clinical Research, Glendale, Arizona
  - AARA Clinical Research, Mesa, Arizona
  - Arthritis and Rheumatism Associates ARA Jonesboro, Jonesboro, Arkansas
  - Clinical Research of West Florida, Clearwater, Florida
  - Omega Research Consultants, DeBary, Florida
  - Suncoast Clinical Research, New Port Richey, Florida
  - Integral Rheumatology And Immunology Specialists, Plantation, Florida
  - Clinical Research of West Florida, Tampa, Florida
  - Clinic of Robert Hozman, Skokie, Illinois
  - Klein And Associates M D P A, Hagerstown, Maryland
  - DM Clinical Research, Brookline, Massachusetts
  - St Paul Rheumatology PA, Eagan, Minnesota
  - Albuquerque Rehabilitation and Rheumatology, Albuquerque, New Mexico
  - Joint and Muscle Research Institute, Charlotte, North Carolina
  - Rheumatology Associates of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Arthritis and Rheumatology Research Institute, Allen, Texas
  - UT Southwestern, Dallas, Texas
  - Naiara Alvarez MD Integrative Rheumatology of South TX, Harlingen, Texas
  - AARA Clinical Research Lone Star Arthritis and Rheumatology, Irving, Texas
  - DM Clinical Research, Tomball, Texas
  - Velocity Clinical Research, Waco, Texas
  - Seattle Rheumatology, Seattle, Washington
- Argentina (6):
  - Instituto Medico De Alta Complejidad (IMAC), Buenos Aires
  - ARCIS Salud SRL Aprillus asistencia e investigacion, Buenos Aires
  - Hospital Militar Central Cir. My. Dr. Cosme Argerich, Buenos Aires
  - Arsema, Ciudad de Buenos Aires
  - Centro Medico Privado de Reumatologia Tucuman, Ciudad de San Miguel de Tucuman
  - MR Medicina Reumatologica, San Fernando
- Australia (5):
  - Ipswich Hospital, Ipswich
  - Rheumatology Research Unit, Maroochydore
  - Queen Elizabeth Hospital, South Woodville
  - Royal North Shore Hospital, St Leonards
  - Royal Darwin Hospital, Tiwi
- Brazil (6):
  - Universidade Federal de Minas Gerais UFMG Faculdade de Medicina, Belo Horizonte
  - LMK Servicos Medicos S S, Porto Alegre
  - Fundacao Faculdade Regional De Medicina S Jose Rio Preto Hospital De Base, São José do Rio Preto
  - BR TRIALS Ensaios Clinicos e Consultoria Ltda, São Paulo
  - CEPIC Centro Paulista de Investigacao Clinica e Servicos Medicos, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Bulgaria (8):
  - UMHAT Kaspela, Plovdiv
  - Multiprofile Hospital for Active Treatment Plovdiv, Plovdiv
  - Diagnostic Consulting Center I Sliven, Sliven
  - Multiprofile Hospital for Active Treatment - MHAT Lyulin EAD, Sofia
  - MC Ekselsior, Sofia
  - Diagnostic-Consultative Center (DCC) Aleksandrovska, Sofia
  - UMHAT St. Ivan Rilski, Sofia
  - ASIMP Rheumatology Centre St Irina EOOD, Sofia
- Canada (7):
  - Eastern Regional Health Authority St Clares Mercy Hospital, St. John's, Newfoundland and Labrador
  - The Waterside Clinic, Orillia, Ontario
  - Womens College Hospital, Toronto, Ontario
  - Alliance Clinical Trials, Waterloo, Ontario
  - Dr Sabeen Anwar Medicine Professional Corporation, Windsor, Ontario
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre de Recherche Musculo Squelettique, Trois-Rivières, Quebec
- China (23):
  - Peking University Third Hospital, Beijing
  - Beijing Tong Ren Hospital Capital Medical University, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Xiangya Hospital Central South University, Changsha
  - West China Hospital Sichuan University, Chengdu
  - Sichuan Provincial Peoples Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - Nanfang Hospital of Southern Medical Hospital, Guangzhou
  - The Affiliated Hospital of Guizhou Medical University, Guiyang
  - Sir Run Run Shaw Hospital Zhejiang University School of Medicine, Hangzhou
  - The First Hospital of Jiaxing, Jiaxing
  - Jinhua municipal central hospital, Jinhua
  - Linyi City People Hospital, Linyi
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Affiliated Hospital of Nantong University, Nantong
  - Pingxiang People's Hospital, Pingxiang
  - Huashan Hospital Fudan University, Shanghai
  - Shanghai skin disease hospital, Shanghai
  - Shenzhen People s Hospital, Shenzhen
  - Second Affiliated Hospital of Soochow University, Suzhou
  - Shanxi Bethune Hospital, Taiyuan
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
- Czechia (9):
  - Revmacentrum MUDr Mostera s r o, Brno
  - Revmatologie s r o, Brno
  - RHEUMA s r o, Břeclav
  - L K N Arthrocentrum, Hlučín
  - CCR Ostrava S R O, Ostrava
  - MUDr Rosypalova s r o, Ostrava
  - FN Motol, Prague
  - Medical Plus S R O, Uherské Hradiště
  - PV Medical S R O, Zlín
- Denmark (6):
  - Aarhus University Hospital, Aarhus N
  - Sydvestjysk Sygehus, Esbjerg
  - Frederiksberg Hospital, Frederiksberg
  - Regionshospitalet Godstrup, Herning
  - Svendborg Hospital Odense University Hospital, Svendborg
  - Vejle Sygehus, Vejle
- Germany (9):
  - Charite - Campus Mitte, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Medizinische Fakultaet Carl Gustav Carus Technische Universitaet Dresden, Dresden
  - Medizinische Fakultaet Der Albert Ludwigs Universitaet Freiburg, Freiburg im Breisgau
  - Hamburger Rheuma Forschungszentrum II, Hamburg
  - Rheumazentrum Ruhrgebiet, Herne
  - Praxis Dr. med. Beate Schwarz - Germany, Langenau
  - Rheumaforschung - Studienambulanz Dr. Wassenberg, Ratingen
  - Universitatsklinikum Tubingen, Tübingen
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Hungary (12):
  - Betegapolo Irgalmas Rend Budai Irgalmasrendi Korhaz, Budapest
  - Revita Kft, Budapest
  - Qualiclinic Kft, Budapest
  - Uno Medical Trials Ltd., Budapest
  - Debreceni Egyetem Reumatologiai Klinika, Debrecen
  - Bekes Varmegyei Kozponti Korhaz Pandy Kalman Tagkorhaz, Gyula
  - Obudai Egeszsegugyi Centrum Kft, Kaposvár
  - Bacs Kiskun Varmegyei Oktatokorhaz, Kecskemét
  - University of Szeged, Szeged
  - Fejer Varmegyei Szent Gyorgy Egyetemi Oktatokorhaz, Székesfehérvár
  - MAV Korhaz es Rendelointezet, Szolnok
  - Vital Medical Center Orvosi es Fogaszati Kozpont, Veszprém
- India (9):
  - Marengo Cims Hospital, Ahmedabad
  - Apollo Hospitals, Bhubaneswar
  - Sushruta Multispeciality Hospital, Hubballi
  - Apollo Multispeciality Hospital Ltd, Kolkata
  - JSS Hospital, Mysuru
  - All India Institute of Medical Sciences, New Delhi
  - Indraprastha Apollo Hospital, New Delhi
  - Fortis Hospital, Noida
  - SIDS (Surat Institute of Digestive Sciences) Hospital and Research Centre, Surat
- Italy (11):
  - A.O. Universitaria Ospedali Riuniti di Ancona, Ancona
  - ASST Spedali Civili Brescia, Brescia
  - Policlinico San Marco, Catania
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Universitaria Luigi Vanvitelli, Napoli
  - IRCCS Policlinico San Matteo, Pavia
  - Universita Degli Studi di Roma Tor Vergata, Roma
  - Fondazione Policlinico Universitario A Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano
  - A O Universitaria Senese Ospedale Santa Maria alle Scotte, Siena
  - Ospedale S. Maria Della Misericordia, Udine
- Japan (13):
  - St. Luke's International Hospital, Chūōku
  - Kansai Medical University Hospital, Hirakata
  - Kita-harima Medical Center, Hyōgo
  - Hospital of the University of Occupational and Enviromental Health, Kitakyushu-shi
  - Nagoya City University Hospital, Nagoya
  - Osaka Metropolitan University Hospital, Osaka
  - Maeshima Rheumatology Clinic, Ōita
  - Sanuki Municipal Hospital, Sanuki
  - Sasebo Chuo Hospital, Sasebo
  - Tohoku University Hospital, Sendai
  - Dokkyo Medical University Hospital, Shimotsuga Gun
  - Kyorin University Hospital, Tokyo
  - Mie University Hospital, Tsu
- Malaysia (6):
  - Hospital Sultanah Bahiyah, Alor Star
  - Hospital Selayang, Batu Caves
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Tuanku Jaafar, Seremban
- Mexico (6):
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, Culiacán
  - Grupo Clinico CATEI, Guadalajara
  - Centro Medico del Angel, Mexicali
  - RM Pharma Specialists, Mexico City
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Centro de Alta Especialidad en Reumatologia e Investigacion, San Luis Potosí City
- Poland (19):
  - Osteo-Medic s.c A. Racewicz, J Supronik, Bialystok
  - Specderm Poznanska sp j, Bialystok
  - ClinicMed Daniluk Nowak Spolka Komandytowa, Bialystok
  - Szpital Uniwersytecki Nr 2 w Bydgoszczy, Bydgoszcz
  - Ambulatorium sp. z o.o., Elblag
  - Centrum Kliniczno Badawcze, Elblag
  - Centrum Medyczne Pratia Gdynia, Gdynia
  - Malopolskie Badania Kliniczne Sp z o o, Krakow
  - Specjalistyczny gabinet dermatologiczny Aplikacyjno Badawczy Marek Brzewski Pawel Brzewski Spolka Cywilna, Krakow
  - Centrum Medyczne All Med, Krakow
  - Pratia MCM Krakow, Krakow
  - Dermed Centrum Medyczne Sp z o o, Lodz
  - Zespol Poradni Specjalistycznych Reumed Filia nr 1, Lublin
  - NZOZ Lecznica MAK MED S C, Nadarzyn
  - MICS Centrum Medyczne Torun, Torun
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Centrum Medyczne Reuma Park, Warsaw
  - DermMedica Sp z o o, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Romania (4):
  - S C Delta Health Care S R L, Bucharest
  - Ecomed Research SRL, Craiova
  - Centrul Medical Unirea, Iași
  - Medaudio Optica S R L, Râmnicu Vâlcea
- Spain (10):
  - Hosp Univ A Coruna, A Coruña
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. de Bellvitge, L'Hospitalet de Llobregat
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp Regional Univ de Malaga, Málaga
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Clinico Univ. de Santiago, Santiago de Compostela
  - Hosp. Virgen Macarena, Seville
  - Hosp. Infanta Luisa, Seville
  - Hosp. Virgen Del Rocio, Seville
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
  - National Taiwan University Hospital Hsin Chu Branch, Taoyuan District
- Thailand (5):
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Saraburi Hospital, Changwat Sara Buri
  - Songklanagarind hospital, Songkhla
- United Kingdom (11):
  - Royal Free London NHS Foundation Trust, Barnet
  - Basingstoke And North Hampshire Hospital, Basingstoke
  - University Hospitals Dorset NHS Foundation Trust, Christchurch
  - Western General Hospital, Edinburgh
  - Glasgow Royal Infirmary, Glasgow
  - Hereford County Hospital, Hereford
  - Forth Valley Royal Hospital, Larbert
  - Haywood Hospital, Staffordshire
  - Torbay Hospital-Devon, Torquay
  - New Cross Hospital, Wolverhampton
  - Betsi Cadwaladr University Health Board BCUHB, Wrexham

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency